CLINICAL TRIAL: NCT01212133
Title: A Post Marketing Surveillance (PMS) Study of Liraglutide in Subjects With Type 2 Diabetes Mellitus in India
Acronym: Lead-In
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3865; U1111-1114-9324 (Other: WHO)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Self-administered subcutaneously (under the skin) once daily at any time, independent of meals, in the abdomen, thigh or upper arm.

SUMMARY:
This study is conducted in Asia. The aim of this study is to evaluate the safety and effectiveness of liraglutide in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes, including newly-diagnosed patients / those already receiving other anti-diabetic medications including GLP-1 analogues, who require treatment with liraglutide according to the clinical judgment of their treating physician
* Subjects who are capable of giving study-specific signed informed consent before any collection of information

Exclusion Criteria:

* Subjects with type 1 diabetes
* Subjects who are or have previously been on liraglutide
* Subjects who have previously been enrolled in the study
* Subjects who are participating in another clinical trial
* Subjects with a hypersensitivity to liraglutide or to any of the excipients (Disodium phosphate dihydrate, propylene glycol, phenol, water for injections)
* Subjects who are pregnant, breast feeding or have the intention of becoming pregnant within the following 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with type 2 diabetes, including newly-diagnosed subjects, who are considered to need treatment with liraglutide are eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 1386 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The number of serious adverse drug reactions (SADRs) during the study period | during 26 weeks of treatment

SECONDARY OUTCOMES:
The number of adverse drug reactions (ADR) during the study period | during 26 weeks of treatment
The number of serious adverse events (SAE) during the study period | during 26 weeks of treatment
Frequency of hypoglycaemic episodes | during 26 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

REFERENCES:
- [Result] Wangnoo SK, Kumar S, Bhattacharyya A, Tripathi S, Akhtar S, Shetty R, Ghosal S. Liraglutide effect and action in diabetes-In (LEAD-In): A prospective observational study assessing safety and effectiveness of liraglutide in patients with type 2 diabetes mellitus treated under routine clinical practice conditions in India. Indian J Endocrinol Metab. 2016 Nov-Dec;20(6):838-845. doi: 10.4103/2230-8210.189232. PMID 27867889
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com